CLINICAL TRIAL: NCT01216098
Title: Impact of Doula Support on Intrapartum Outcomes for Women Undergoing a Vaginal Birth After Cesarean (VBAC)
Brief Title: Impact of Doula Support on Childbirth Outcomes for Women Undergoing a Vaginal Birth After Cesarean (VBAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Provincial Health Services Authority (PHSA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H10-01551
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Cesarean
Keywords: Intrapartum; Clinical trial; Perinatal; Doula; VBAC; Perinatal Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm - D (Experimental): Experimental arm - Women randomized to this arm will receive doula support alongside standard care.
  Interventions: Behavioral: Doula support
- No intervention - ND (No Intervention): No intervention - Women randomized to this arm will receive standard care alone.

INTERVENTIONS:
Behavioral: Doula support — A doula is a paraprofessional who provides continuous emotional and physical support to women and their families during the intrapartum period.
  Arms: Experimental arm - D

SUMMARY:
The purpose of this study is to evaluate the impact of doula support on childbirth outcomes of women who are eligible for and attempting to have a Vaginal Birth After Cesarean (VBAC). Doulas are paraprofessionals who provide women with continuous physical and emotional support throughout the course of labour. They also conduct home visits in the prenatal and postpartum periods in order to provide women with information on childbirth-related topics and breastfeeding support. They do not perform clinical tasks. Their value lies in the psycho-social care that they provide. It is hypothesized that women who receive doula support alongside standard care will have a lower rate of epidural analgesia use and greater cervical dilation at time of epidural administration, as compared to those who receive standard care alone.

DETAILED DESCRIPTION:
A two-armed randomized controlled trial will be conducted at BC Women's Hospital. The experimental group will receive both standard clinical care and doula support. The control group will receive standard clinical care without doula support. The main outcomes being looked at are use of epidural analgesia and cervical dilation at time of epidural administration. These outcomes have been chosen because of the association between the use of epidural analgesia and both a prolonged length of labour and the need for assisted deliveries (i.e. forceps assisted deliveries, vacuum assisted deliveries, and cesarean births). If it is found that providing doula support for women who are eligible for and attempting to have a VBAC reduces or delays the use of epidural analgesia, then it could be hypothesized that doula support for this population may also shorten the length of labour and reduce the need for assisted deliveries, thereby justifying ongoing research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Women who have had at least one prior cesarean birth, are eligible for VBAC, and plan to attempt a VBAC after counseling at the Best Birth Clinic.
* Singleton gestation.
* Cephalic presentation.
* Term gestation (37-42 weeks at time of delivery).

Exclusion Criteria:

* Women who have a pre-existing medical condition that would be an indication for an elective cesarean birth.
* Women who plan to privately hire a doula regardless of placement in either arm of the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Use of epidural analgesia and cervical dilation at time of epidural administration.
  The main outcomes being looked at are use of epidural analgesia and cervical dilation at time of epidural administration. This information will be recorded in the patient charts during the intrapartum period and collected from these charts at a later date by a research assistant.

SECONDARY OUTCOMES:
Cervical dilation at time of epidural administration
  The following secondary outcomes will be measured:
  * Use of nitrous oxide analgesia during labour.
  * Use of narcotic analgesia during labour (type and amount).
  * Number of visits to the assessment room before admission.
  * Mode of delivery (cesarean section, spontaneous vaginal, or forceps/vacuum).
  * Indication(s) for repeat cesarean (if applicable).
  * Length of time between admission and the start of active pushing.
  * Length of time between the start of active pushing and delivery.
  * Length of time between delivery and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Janssen, BSN, MPH, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://www.powertopush.ca/info-for-professionals/more-about-the-campaign/